CLINICAL TRIAL: NCT01875445
Title: A Double-Blind, Placebo-Controlled Study of Inositol in Trichotillomania
Brief Title: Inositol in Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013InositolTTM
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania; Hair Pulling
Keywords: Inositol; Trichotillomania; Hair Pulling; Impulse Control Disorder
MeSH Terms: conditions — Trichotillomania; Disruptive, Impulse Control, and Conduct Disorders | interventions — Inositol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matched dosage of inositol daily.
  Interventions: Drug: Placebo
- Inositol (Active Comparator): Powder form, 2g TID up to 6g TID
  Interventions: Drug: Inositol

INTERVENTIONS:
Drug: Inositol — Taken as 2g of powder TID for 2 weeks, then 4g of powder TID for 2 weeks and then 6g of powder TID for the remainder of the study.
  Other Names: Inositol Powder
  Arms: Inositol
Drug: Placebo — Taken as 2g of powder TID for 2 weeks, then 4g of powder TID for 2 weeks and then 6g of powder TID for the remainder of the study.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of inositol for the treatment of compulsive hair pulling, also known as trichotillomania. Inositol is used for diabetic nerve pain, panic disorder, high cholesterol, insomnia, cancer, depression, schizophrenia, Alzheimer's disease, attention deficit-hyperactivity disorder (ADHD), autism, promoting hair growth, a skin disorder called psoriasis, and treating side effects of medical treatment with some medications, including lithium. The hypothesis to be tested is that Inositol will be effective and well tolerated in patients with trichotillomania compared to placebo. The proposed study will provide needed data on the treatment of the disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
Pathological hair-pulling, trichotillomania, has been defined as repetitive, intentionally performed pulling that causes noticeable hair loss and results in clinically significant distress or functional impairment (1). Trichotillomania appears relatively common with an estimated prevalence between 1-3% (2). Data on the pharmacological treatment of trichotillomania is limited to case reports and conflicting double-blind studies of serotonin reuptake inhibitors (3).

Inositol is used for diabetic nerve pain, panic disorder, high cholesterol, insomnia, cancer, depression, schizophrenia, Alzheimer's disease, attention deficit-hyperactivity disorder (ADHD), autism, promoting hair growth, a skin disorder called psoriasis, and treating side effects of medical treatment with some medications, including lithium. A small study (n=3) found that subject's showed improvement while taking Inositol in both trichotillomania and pathological skin picking (4). This suggests that Inositol might be effective in treating a large sample of subjects with trichotillomania and it also suggests that it may be effective for impulse control disorders in general. Inositol has also been shown to be effective in treating obsessive compulsive disorder and showed significantly lower scores on the Yale-Brown Obsessive Compulsive Scale (5). Both studies indicate the effectiveness of Inositol in treating impulsivity and compulsivity in subjects. There is no medication approved by the Food and Drug Administration for trichotillomania. Inositol represents a potentially safe and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Trichotillomania (TTM) as the primary psychiatric diagnosis
3. Women's participation required negative results on a beta-human chorionic gonadotropin pregnancy test and stable use of a medically accepted form of contraception.
4. Signed informed consent before entry into the study.

Exclusion Criteria:

1. Unstable medical illness or clinically significant abnormalities on laboratory tests or physical examination at screening visit
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. A need for medication other than ecopipam with possible psychotropic effects
4. Lifetime history of bipolar disorder type I or II, dementia, or schizophrenia as determined by the Structured Clinical Interview for DSM-IV
5. Current (past 12-months) DSM-IV substance abuse or dependence
6. Positive urine drug screen at screening
7. Initiation of cognitive behavior therapy within 3 months prior to study baseline
8. Baseline score of ≥17 on the Hamilton Depression Rating Scale (17-item HDRS
9. Any suicidality based on clinical interview
10. History of head injury or neurological disorder (such as seizures)
11. Any history of psychiatric hospitalization in the past year
12. Any history of a suicide attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD,JD,MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Inositol
Started | 19 | 19
Completed | 12 | 19
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Inositol | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (12.2) | 28.0 (11.4) | 28.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 17 | 18 | 35
  Race/Ethnicity: African American | 2 | 0 | 2
  Race/Ethnicity: Latino/Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
National Institute of Mental Health Trichotillomania Severity Scale [Mean (Standard Deviation); unit: units on a scale] — A standard clinician administered scale to assess trichotillomania symptom severity. Scale range of 0-25. Higher scores indicate greater severity.
  units on a scale | 11.6 (3.4) | 12.9 (3.7) | 12.3 (3.6)
Massachusetts General Hospital Hairpulling Scale [Mean (Standard Deviation); unit: units on a scale] — A standard self-report scale to assess trichotillomania symptom severity. Scale range of 0-28. Higher scores indicate greater severity.
  units on a scale | 17.9 (3.3) | 18.8 (4.2) | 18.4 (3.8)
The Clinical Global Impressions Scale-Severity [Mean (Standard Deviation); unit: units on a scale] — A clinician rating of disorder severity with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.2 (.5) | 4.5 (.6) | 4.4 (.6)

OUTCOME MEASURES:

1. Primary Outcome: The National Institute of Mental Health Trichotillomania Symptom Severity Scale (NIMH-TSS)
Description: The entire study for an individual subject will last 10 weeks. Every 2 weeks the subject will take the NIMH-TSS for the duration of the 10 weeks, but only baseline and final values will be used for general final outcome assessment. The scale itself asses severity of hair pulling.
Time Frame: Once every two weeks for the 10 weeks of the study
Population: Last observation carried forward for general means.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Inositol
Number analyzed (Participants) | 19 | 19
units on a scale | 8.4 (5.5) | 8.4 (5.1)

2. Secondary Outcome: The Massachusetts General Hospital (MGH) Hairpulling Scale
Description: The entire study for an individual subject will last 10 weeks. Every 2 weeks the subject will take the MGH Hairpulling Scale for the duration of the 10 weeks, baseline and final visits will be use for general final outcome assessment. The scale itself asses severity of hair pulling.
Time Frame: Once every two weeks for the 10 weeks of the study
Population: Last observation carried forwards for general averages.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Inositol
Number analyzed (Participants) | 19 | 19
units on a scale | 14.5 (5.1) | 13.2 (6.8)

ADVERSE EVENTS:
Arm/Group | Placebo | Inositol
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 4/19 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Inositol (N=19)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Subject reported an ectopic pregnancy during the study. This was a possible side effect of the subject's birth control medication, and was thus unlikely to be related to the inositol treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Inositol (N=19)
Nausea/Upset Stomach (Gastrointestinal disorders) | 2 (3) | 4 (6) — Mild severity.
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) — Mild severity.
Headache (General disorders) | 2 (2) | 2 (2) — Mild severity.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No